CLINICAL TRIAL: NCT07264608
Title: Comparison of 4-Point Transversus Abdominis Plane Block and Combined Bilateral Rectus Sheath-Oblique Subcostal TAP Block on Quality of Recovery After Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: 4-Point TAP Block vs. Combined RSB-OSTAP Block for Recovery After Laparoscopic Cholecystectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Esma Karaarslan, Medical Doctor (MD), Department of Anesthesiology and Reanimation, Konya City Hospital, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4TAB-RSB
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain; Quality of Recovery
Keywords: Quality of recovery; TAP block; Rectus sheath block; OSTAP block; Laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4-Point TAP (4QTAP) Group (Experimental): An ultrasound-guided 4-point transversus abdominis plane block will be performed at two subcostal and two lateral anatomical sites. A total of 40 mL of 0.25% bupivacaine will be administered, with 10 mL injected at each point
  Interventions: Procedure: 4-Point TAP (4QTAP) Group
- RSB + OSTAP Group (Active Comparator): A combined bilateral rectus sheath block and bilateral oblique subcostal TAP block will be performed under ultrasound guidance. Four injection points (two RSB + two OSTAP) will be used, and a total of 40 mL of 0.25% bupivacaine will be administered, with 10 mL injected at each point.
  Interventions: Procedure: RSB + OSTAP Group

INTERVENTIONS:
Procedure: 4-Point TAP (4QTAP) Group — 4-Point TAP (4QTAP) Group: Ultrasound-guided 4-point transversus abdominis plane block will be performed at two subcostal and two lateral injection points. A total of 40 mL of 0.25% bupivacaine will be administered (10 mL at each point).
  Arms: 4-Point TAP (4QTAP) Group
Procedure: RSB + OSTAP Group — RSB + OSTAP Group:
  Ultrasound-guided bilateral rectus sheath block (two injection points) combined with bilateral oblique subcostal TAP block (two injection points) will be performed. A total of 40 mL of 0.25% bupivacaine will be administered (10 mL at each point).
  Arms: RSB + OSTAP Group

SUMMARY:
Laparoscopic cholecystectomy is a common keyhole surgery to remove the gallbladder. Although the cuts are small, patients can still have significant pain and nausea after the operation, which may delay recovery and discharge. To improve comfort, doctors often use ultrasound-guided abdominal nerve blocks as part of multimodal pain management.

In this single-center, randomized controlled trial, adult patients scheduled for elective laparoscopic cholecystectomy will receive standard general anesthesia and be randomly assigned to one of two routinely used block techniques at the end of surgery: (1) a 4-point transversus abdominis plane (TAP) block, or (2) a combined bilateral rectus sheath block plus oblique subcostal TAP block. Both techniques are performed under ultrasound guidance while the patient is still asleep.

The main aim of the study is to compare the quality of recovery on the first day after surgery between the two groups, using a short questionnaire (QoR-15). Secondary aims are to compare pain scores, the need for additional pain medicine, and the frequency of postoperative nausea and vomiting between the groups during the first 24 hours. All other aspects of anesthesia and surgical care will follow standard hospital practice. Participation is not expected to add significant risk beyond that of routine anesthesia and surgery, as both block techniques are already commonly used in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-65 years

ASA physical status I-II

Scheduled for elective laparoscopic cholecystectomy

Ability to understand the study and provide written informed consent

Exclusion Criteria:

Allergy or hypersensitivity to local anesthetics or study medications

Coagulopathy, anticoagulant therapy, or local infection at block site

Severe pulmonary disease (severe COPD, uncontrolled asthma, respiratory failure)

NYHA class III-IV heart failure

History of thoracic or abdominal surgery affecting block area

Chronic pain syndrome or regular opioid/analgesic use

Morbid obesity (BMI > 35 kg/m²)

Pregnancy or breastfeeding

Cognitive impairment preventing cooperation

Conversion to open cholecystectomy

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery score (QoR-15) | 24 hours
  The Quality of Recovery-15 (QoR-15) questionnaire will be used to assess postoperative recovery quality at 24 hours after surgery.
  The QoR-15 scale ranges from 0 to 150 points, with higher scores indicating better recovery quality.

SECONDARY OUTCOMES:
Postoperative pain score (VAS) | 30 minutes, 2 hours, 8 hours, and 24 hours after surgery.
  Postoperative pain intensity will be evaluated using the Visual Analog Scale (VAS) at predefined time points.
  The VAS scale ranges from 0 to 10, where 0 represents no pain and 10 represents the worst imaginable pain. Higher scores indicate worse pain.
Incidence of postoperative nausea and vomiting (PONV) | First 24 hours postoperative.
  Presence and severity of nausea (0-3 scale) and vomiting episodes (0-3 scale).
Antiemetic requirement | First 24 hours postoperative.
  Number of patients requiring intravenous ondansetron based on nausea (≥2) or vomiting (≥1).

CONTACTS AND LOCATIONS:
Overall Officials: Esma karaarslan, MD, Principal Investigator — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No